CLINICAL TRIAL: NCT00934024
Title: Impact of Varenicline on Blood-Oxygen-Level Dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Activation on Smokers (GRAND)
Brief Title: Impact of Varenicline on Blood-Oxygen-Level Dependent (BOLD) Functional Magnetic Resonance Imaging (fMRI) Activation on Smokers
Acronym: GRAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR#18521
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Nicotine Dependence
Keywords: nicotine dependence; tobacco; smoking
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Varenicline

ARMS (2):
- Abstinent (Other): All participants received varenicline. A priori determined analysis was between participants who quit smoking and those who continued to smoke.
  This arm was abstinent after 5 weeks of varenicline treatment..
  Interventions: Drug: varenicline
- Non-abstinent (Other): All participants received varenicline. A priori determined analysis was between participants who quit smoking and those who continued to smoke.
  This arm was participants who continued to smoke after 5 weeks of varenicline treatment.
  Interventions: Drug: varenicline

INTERVENTIONS:
Drug: varenicline — Participants will be treated with a standard course of varenicline, 0.5 mg 1 tablet every day for 3 days, then 0.5 mg 1 tab twice a day for four days, and 1 mg 1 tablet twice a day for three months.
  Other Names: Chantix

SUMMARY:
The purpose of this study is to evaluate the impact of varenicline treatment on cue induced craving to smoking using brain imaging. The investigators hypothesize that participants will report reduced urges to smoke and will have less activation in parts of the brain associated with craving.

DETAILED DESCRIPTION:
Treatment with varenicline reduces overall subjective cigarette craving and smoking reward in nicotine-dependent smokers. This preliminary study will explore the impact of varenicline treatment on smoking cue-induced craving and associated regional brain activation using BOLD fMRI. Twenty healthy smokers (10 males, 10 females) will undergo two BOLD fMRI scans with the presentation of smoking-related and neutral cues at baseline and after five weeks of treatment with open-label varenicline. The investigators hypothesize that participants will report reduced urges to smoke on the Questionnaire of Smoking Urges-Brief and have less activation of the brain areas associated with craving during the fMRI after 5 weeks of varenicline and smoking cessation counseling compared to the baseline scan.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 - 60 treatment-seeking right handed smokers.
2. Meet criteria for primary nicotine dependence confirmed by FTND and smoked at least 70% of days in the last 30 days prior to assessment.
3. General good health confirmed by history & physical.
4. Able to read and understand questionnaires and informed consent.
5. Motivated to quit, willing to set a target quit date (TQD) and abstain from smoking after TDQ.
6. Participants must have a negative urine drug screen (UDS) and pregnancy test prior to imaging sessions and beginning varenicline treatment.
7. Female participants will use a reliable method of birth control throughout the study.
8. Demonstrate subjective response to cues in a laboratory cue reactivity session.

Exclusion Criteria:

1. Currently meets DSM-IV criteria for any other psychoactive substance dependence disorder except nicotine dependence.
2. Any psychoactive substance abuse within the last 30 days as evidenced by subject report or urine drug screen.
3. Use of other tobacco products.
4. Current use of nicotine replacement therapy, bupropion, or other smoking cessation treatment.
5. Previous failed attempt on varenicline.
6. Meets DSM-IV criteria for current axis I disorders of major depression, panic disorder, obsessive compulsive disorder, post-traumatic stress syndrome, bipolar affective disorder, schizophrenia, or any other psychotic disorder or organic mental disorder.
7. Current suicidal ideation with plan or homicidal ideation.
8. Need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications which could potentially interfere with fMRI.
9. Clinically significant medical problems that would impair participation or limit ability to participate in scan.
10. Sexually active females of child-bearing potential who are pregnant, nursing, or who are not using a reliable form of birth control.
11. Has current charges pending for a violent crime (not including DUI related offenses).
12. Persons with ferrous metal implants or pacemaker since fMRI will be used.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Hartwell, M.D., Principal Investigator — Medical Universtiy of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Right-handed nicotine dependent cigarette smokers between 21 and 60 years of age were recruited via community and internet advertisements. Recruitment took place between 2009 and 2011.
Pre-assignment Details: All participants received open-label varenicline. Participants data was anaylzed in two groups- abstinent and non-abstinent participants.
Groups:
- Non-abstinent: All participants received varenicline. A priori determined analysis was between participants who quit smoking and those who continued to smoke.
  This arm was people who continued to smoke after 5 weeks of varenicline treatment.
Period: Overall Study
Arm/Group | Abstinent | Non-abstinent
Started | 10 | 11
Completed | 10 | 6
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abstinent | Non-Abstinent | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.8 (13.07) | 35.55 (11.72) | 30.18 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] | 20.45 (5.83) | 17.27 (4.29) | 18.86 (5.06)

OUTCOME MEASURES:

1. Primary Outcome: Change in Post-Resist Craving
Description: Change in Post-resist task craving between Scan 1, pre-medication, and Scan 2, post- medication, as measured on a 0-10 Likert scale. The Within Sessions Rating scale (Range 0-10) measures craving with 0 indicating Not at All and 10 indicating Extremely. Change scores were calculate by subtracting the craving score immediately following the pre-medication scan from the craving score immediately following the post-medication scan.
Time Frame: 5 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Abstinent: All participants received varenicline. A priori determined analysis was between participants who quit smoking and those who continued to smoke.
  This arm was abstinent after 5 weeks of varenicline treatment..
  varenicline: Participants will be treated with a standard course of varenicline, 0.5 mg 1 tablet every day for 3 days, then 0.5 mg 1 tab twice a day for four days, and 1 mg 1 tablet twice a day for three months.
- Non-abstinent: All participants received varenicline. A priori determined analysis was between participants who quit smoking and those who continued to smoke.
  This arm was participants who continued to smoke after 5 weeks of varenicline treatment.
  varenicline: Participants will be treated with a standard course of varenicline, 0.5 mg 1 tablet every day for 3 days, then 0.5 mg 1 tab twice a day for four days, and 1 mg 1 tablet twice a day for three months.
Arm/Group | Abstinent | Non-abstinent
Number analyzed (Participants) | 10 | 6
units on a scale | 6 (1.41) | 3.6 (1.14)

ADVERSE EVENTS:
Time Frame: AE's were collected over 5 weeks post medication administration.
Groups:
- All Participants: All participants received varenicline. A priori determined analysis was between participants who quit smoking and those who continued to smoke.
  Adverse events are reported for the total of all participants. Since all patients received medication, DSMB reports were made in aggregate and are reported as such here.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 16/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=21)
Localized rash (Skin and subcutaneous tissue disorders) | 1 (1)
Head, Eyes, Ears, Nose, Throat (General disorders) | 8 (8) — Sore throat, difficulty swallowing, headache, nasal congestion, lightheaded, mouth tenderness, tinnitus, URI
Gastrointestinal (Gastrointestinal disorders) | 10 (10) — Nausea, diarrhea, increased belching, constipation, GI illness, vomiting, reflux, loose stools
Sleep Related (General disorders) | 11 (11) — Insomnia, drowsiness, vivid dreams, talking in sleep
Psychiatric (Psychiatric disorders) | 3 (3) — Irritability, Increased sadness
Peripheral vascular (Vascular disorders) | 2 (2) — Ankle swelling, hand swelling
General (General disorders) | 5 (5) — Fever, Minimal weight gain, Increased appetite

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes